CLINICAL TRIAL: NCT02882672
Title: Exercise-based Cardiac Rehabilitation
Brief Title: Changes in Adiponectin and Cardiovascular Disease Risk Factors in Overweight Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Isfahan (Other)
Responsible Party: Principal Investigator, Prof.Mehdi Kargarfard, Professor Mehdi Kargarfard, University of Isfahan
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201527898IR
Record Dates: First submitted 2016-08-12; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Exercise; Cardiac Myosins; Patients
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): experimental group did 8 weeks exercise training
  Interventions: Other: Experimental
- Control (Experimental): Control group did not do any exercise training.
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — Doing exercise at 60-85% of maximal heart rate, lasted 45-60 minutes and included a 10-minute warm-up, 40 minutes of aerobic exercises, consisting of stationary cycling, walking and/or jogging
  Arms: Experimental
Other: Control — They did not do ant exercise training during 8 weeks.
  Arms: Control

SUMMARY:
This study aimed to determine if eight-weeks of exercise-based cardiac rehabilitation could improve adiponectin and cardiovascular disease risk factors in overweight coronary heart disease patients. Patients were included in the study if: they were approved to do so following a physical, physiological and psychological test; did not take part in regular physical activity; had stable heart failure for at least 3 months. Exclusion criteria included: a history of surgery within the preceding 4 months; had an unstable angina, acute phase of myocardial infarction, and/or unstable arrhythmia; had obstructive cardiomyopathy, exercise-induced ischemia or arrhythmias, uncontrolled arrhythmias, resting blood pressure more than 200/120 millimeters mercury, aortic stenosis, and/or peripheral artery disease; exercise limitations due to neuromuscular and/or musculoskeletal disease; had any health problems that prevented maximum effort on the treadmill test. Target population included of all patients with a history of myocardial infarction and diagnosis of congestive heart failure who were referred to Isfahan Cardiovascular Research Centre. 60overweight coronary heart disease patients were randomly assigned to either an eight-week, three times weekly exercise group (n=30), or a non-exercising control group (n=30). Exercise sessions took place at 60-85% of maximal heart rate, lasted 45-60 minutes and included a 10-minute warm-up, 40 minutes of aerobic exercises, consisting of stationary cycling, walking and/or jogging, flexibility, balance exercises, and weight-bearing activity and a 10-minute cool-down.

ELIGIBILITY:
Inclusion Criteria:

* they were approved to do so following a physical, physiological and psychological test; resided and worked in the city of Isfahan; did not take part in regular physical activity; had stable heart failure for at least 3 months.

Exclusion Criteria:

* a history of surgery within the preceding 4 months
* had an unstable angina, acute phase of myocardial infarction (MI), and/or unstable arrhythmia
* had obstructive cardiomyopathy, exercise-induced ischemia or arrhythmias, uncontrolled arrhythmias, resting blood pressure more than 200/120 millimeters mercury (mmHg), aortic stenosis, and/or peripheral artery disease
* exercise limitations due to neuromuscular and/or musculoskeletal disease, such as any type of orthopedic, low back pain, bone fracture of less than 6 months
* uncontrolled systemic disease, such as DM; were 75 years or older
* had any health problems that prevented maximum effort on the treadmill test
* unable to answer the screening questionnaires assessing depression and anxiety.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-01; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Effect of Exercise-based cardiac rehabilitation on Serum levels of adiponectin was measured by ELISA method | up to 8 weeks
  Exercise sessions took place at 60-85% of maximal heart rate, lasted 45-60 minutes.
Effect of Exercise-based cardiac rehabilitation on lipids was measured by ELISA method | up to 8 weeks

SECONDARY OUTCOMES:
Effect of Exercise-based cardiac rehabilitation on weight was measured | up to 8 weks
Effect of Exercise-based cardiac rehabilitation on height was measured | up to 8 weks

IPD SHARING:
Plan to Share IPD: No